CLINICAL TRIAL: NCT03145662
Title: Cutting Balloon vs. High Pressure Balloon for the Treatment of AV Graft Stenosis
Brief Title: High Pressure Balloon vs Cutting Balloon
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Resources
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Munier Nazzal, M.S. M.D, MD, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPB vs CB
Record Dates: First submitted 2017-03-24; First posted 2017-05-09 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Intervention Model Description: randomization to either high pressure balloon or cutting balloon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- high pressure balloon (Active Comparator): randomized to have dialysis fistula or AV graft treated with high pressure balloon
  Interventions: Device: high pressure balloon
- cutting balloon (Active Comparator): randomized to have dialysis fistula or AV graft treated with cutting balloon
  Interventions: Device: cutting balloon

INTERVENTIONS:
Device: high pressure balloon — high pressure balloon will be used to treat stenosis
  Arms: high pressure balloon
Device: cutting balloon — cutting balloon will be used to treat stenosis
  Arms: cutting balloon

SUMMARY:
Patients suspected of having AV access stenosis will be referred to the Division of Vascular and Endovascular Surgery by the dialysis center. Patients with signs of AV access failure who are found to have significant stenosis (more than 50%) at the venous end of the anastomosis will then be randomized to either high pressure balloon (Conquest) or to a cutting balloon (Boston scientific Balloon). Angiograms will then be performed before and after intervention.

DETAILED DESCRIPTION:
Patients suspected of having AV access stenosis will be referred to the Division of Vascular and Endovascular Surgery by the dialysis center. Patients with signs of AV access failure who are found to have significant stenosis (more than 50%) at the venous end of the anastomosis will then be randomized to either high pressure balloon (Conquest) or to a cutting balloon (Boston scientific Balloon). Angiograms will then be performed before and after intervention.

Data will be collected from standard of care visit, including physician visits and ultrasounds. Follow up will be based on the function of the AV access, dialysis center criteria and/or standard of care ultrasound results: including venous pressure of the AV access, difficult cannulation, urea recirculation, and change in character and sound of the AV access (thrill/bruit), which are standard of care assessment at a dialysis center. All patient data sheets will be kept in a study binder and locked in the research room. Randomization will be performed with a computer program.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. AV fistula or graft
3. Undergoing weekly hemodialysis
4. Patients must agree to the terms of the study and sign an informed Consent

Exclusion Criteria:

1. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Stenosis Rate | 2 years
  days of stenosis free period

CONTACTS AND LOCATIONS:
Locations (1):
- UTMC, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No